CLINICAL TRIAL: NCT04243811
Title: Efficacy of Low Level Laser Therapy in the Management of Injection Pain During Supraperiosteal Anesthesia in Children: A Randomize Clinical Trial
Brief Title: Efficacy of Low Level Laser Therapy on İnjection Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the technical problem in the laser device,it has not started.
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Sinem yildirim, Assist. Prof. Dr., Okan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018/47
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Pediatric Anesthesia; Low Level Laser Theraphy
Keywords: pediatric patient; injection pain; lllt
MeSH Terms: interventions — Lasers, Semiconductor; Anesthesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser group (Experimental): local anesthesia applyed with 940 nm diode laser
  Interventions: Device: Diode Laser
- conventional group (Active Comparator): local anesthesia applyed with topical anesthesia
  Interventions: Other: topical anesthesia

INTERVENTIONS:
Device: Diode Laser — LLLT with dental needle for local anesthesia during dental treatment
  Arms: laser group
Other: topical anesthesia — topical anesthesia with dental needle for local anesthesia during dental treatment
  Arms: conventional group

SUMMARY:
The purpose of this study was to compare the pain during needle insertion and injection in supraperiosteal anesthesia with either topical anesthesia (control) or LLTT (experimental).

ELIGIBILITY:
Inclusion Criteria:

In need of treatment of right and left molar teeth of maxilla,

* Does not have any systemic disorder,
* High level of communication that can provide logical answers to the questions we ask
* With parental consent,
* Volunteers who want to participate in the research
* 6-12 years old patients who are compatible with routine dental treatments in the pediatric clinic

Exclusion Criteria:

* No need for treatment of right and left molar teeth of maxilla,
* Has a systemic condition
* Low level of communication that cannot provide reasonable answers to the questions we ask
* Without parental consent
* Do not want to participate voluntarily in the research
* Do not attend a check-in
* Patients not in the 6-12 age group

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
Wong-Baker Faces Pain Rating Scale (PRS) | 1 year
  The PRS measures the unpleasantness or affective dimension of a child's pain experience and is used in children aged 3-17 years old. The PRS consists of a set of cartoon faces with varying facial expressions ranging from a smile/laughter to tears, and each child is asked to select the facial expression that best represents his/her experience of discomfort. Each face has a numerical value ranging from 0 (smiling face, "no hurt") to 5 (crying/screaming face, "hurts worst").
Face, Legg, Cry, Consolability Scale (FLACC) | 1 year
  The scale comprised the following parameters: (1) Face, (2) Legs, (3) Activity, (4) Cry, and (5) Consolability. Each of the five categories is scored from 0-2, which results in a minimum total score of 0 and maximumof 10. According to this scale: 0=Relaxed and comfortable (no pain); 1-3=Mild discomfort; 4-6=Moderate pain; and 7-10=Severe discomfort or pain [Willis et al., 2003]. Behavioural parameters were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Okan University Faculty of Dentistry, Istanbul, Turkey (Türkiye)